CLINICAL TRIAL: NCT04597892
Title: Efficacy of Point-of-care Creatinine Assays in Patients With eGFR <30ml/Min/1.73m2 in the Setting of Elective Procedures With Intravascular Iodinated Contrast
Brief Title: Efficacy of Point-Of-Care Creatinine Assays in Patients With eGFR <30 Receiving Intravascular Contrast
Acronym: EPIC
Status: Withdrawn | Type: Observational
Why Stopped: delay
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL.MUMC.AMACINGrp.3
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Renal Insufficiency; Acute Kidney Injury; Contrast-induced Nephropathy
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum creatinine assay — point-of-care and standard laboratory assay of serum creatinine

SUMMARY:
Point-of-care (POC) creatinine devices allow rapid measurement of creatinine levels and calculation of estimated glomerular filtration rate (eGFR) which give an indication of renal function. The focus of this assessment is to validate POC measurements to assess kidney function before intravascular iodinated contrast administration in patients with severe renal insufficiency (eGFR < 30 ml/min/1.73m2). It will be evaluated whether discrepancies between POC measurement values and values obtained from standard laboratory assays lie within an acceptable range using Bland-Altman analysis.

DETAILED DESCRIPTION:
Measurement of creatinine to determine eGFR before intravascular iodinated contrast administration is indicated to assess whether a patient is at risk of contrast-induced acute kidney injury (AKI). For patients with reduced eGFR intravenous hydration can be offered before the scan to reduce the risk of AKI. If no recent eGFR measurement is available, contrast procedures could be cancelled and rescheduled while a creatinine test is processed in the laboratory. Using POC creatinine tests before contrast-enhanced procedures could minimise the risk of kidney injury, and may reduce the number of cancelled scans. The question is whether POC creatinine assay is accurate and beneficial in this setting compared to the standard laboratory assay.

The i-STAT Alinity POC creatinine device is one of three devices which calculate estimated glomerular filtration rate (eGFR) recommended in clinical practice guidelines to assess kidney function to guide decisions on the use of intravascular iodinated contrast in adults. In the study, i-STAT Alinity POC measurements of creatinine will be performed using already available blood samples of patients with estimated eGFR<30 ml/min/1.73m2 and mean difference between eGFR and serum creatinine measurements using POC and standard laboratory assays will be calculated. Results will be used to evaluate the agreement between of POC and laboratory assays on risk stratification (i.e., the percentage of patients with eGFR<30 according to both laboratory and POC assays) and post-contrast acute kidney injury (AKI; i.e., the percentage of patients with post-contrast acute kidney injury according to both laboratory and POC assays). Finally, the number of elective procedures which are delayed (including delayed planning) or cancelled because a serum creatinine assay is required and unavailable will be prospectively evaluated for Maastricht UMC+ in this study.

ELIGIBILITY:
Inclusion Criteria:

* Standard care venous blood samples for which eGFR measurement at Maastricht UMC+ Central Diagnostic Laboratory results in a value below 30 ml/min/1.73m2 (including all standard care venous blood samples from patients with GFR <30 ml/min/1.73m2 referred for an elective procedure with intravascular iodinated contrast at Maastricht UMC+)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Standard care venous blood samples for which eGFR measurement at Maastricht UMC+ Central Diagnostic Laboratory have resulted in a value below 30 ml/min/1.73m2 (including all standard care venous blood samples from patients with GFR <30 ml/min/1.73m2 referred for an elective procedure with intravascular iodinated contrast at Maastricht UMC+) will be used in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2097-05-01 (Estimated); Primary Completion 2099-03-01 (Estimated); Study Completion 2099-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean difference between eGFR and serum creatinine measurements using POC and standard laboratory assays | 6 months
  with 95% limits of agreement (based on the standard deviation of the individual between-method differences).

SECONDARY OUTCOMES:
Agreement risk stratification. | 6 months
  percentage of patients classified as eGFR <30 by both POC and standard laboratory assays
Agreement post-contrast acute kidney injury. | 6 months
  percentage of patients with post-contrast AKI according to both POC and standard laboratory assays

OTHER OUTCOMES:
Delayed/cancelled procedures. | 6 months
  The percentage of elective procedures which are delayed (including delayed planning) or cancelled because a serum creatinine assay is required and unavailable will be prospectively evaluated for Maastricht UMC+ in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No